CLINICAL TRIAL: NCT02665611
Title: The Effect of Remote Monitoring and Support for Patients Suffering From Schizophrenia, Schizoaffective or Bipolar Disorder on Adherence to Treatment
Brief Title: Remote Monitoring and Support for Patients With Schizophrenia, Schizoaffective or Bipolar Disorder on Adherence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assuta Hospital Systems (Other)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2124-15-SMC
Record Dates: First submitted 2016-01-18; First posted 2016-01-28 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder | interventions — Methods; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention group (Experimental): intervention for improvement of treatment adherence "Intervention group"- This group will be followed by the "MOMA" call center (By the MOMA nures every couple weeks and by the study coordinatore and the treating Doctor at special "visits" as the study required.) The group will be monitored according to number of parameters, including treatment Adherence.
  Interventions: Behavioral: intervention for improvement of adherence
- control group (Experimental): treatment as usual Control group- Treatment will continue as usual by the Doctor.(This group will allso be followed by the Study Coordinator at the same "visits" as the "Intervention group".The group will be monitored according to number of parameters, including treatment Adherence.
  Interventions: Behavioral: treatment as usual

INTERVENTIONS:
Behavioral: intervention for improvement of adherence — intervention for improvement of adherence
  Arms: intervention group
Behavioral: treatment as usual — The control group will be treated according to the usual stadard of care.
  Arms: control group

SUMMARY:
Moma call center will provide unique service -Remote monitoring and support for mental health patients .The aim of this reserch is reducing hospitalization and improve adherence, by reaching out and there for monitoring very closely .

DETAILED DESCRIPTION:
"Moma" call center is a result of collaboration between Maccabi Health Services and The Gertner Institute of Epidemiology and Health Policy Research. The call center provides remote continuous monitoring and support for patients with chronic illnesses, and has been found useful for improvement in treatment adherence and other clinical measures in patients with diabetes and CHF.

The current project focuses on patients diagnosed with schizophrenia, schizoaffective disorder and bipolar disorder. Patients that suffer from these disorders are prone to low adherence and are at risk for discontinuation of treatment and frequent relapses.

The advantages of the "Moma" call-center include high availability, reaching out, collaboration between treatment centers and agents, and continuous remote monitoring. We hypothesize that these factors will enable improvement of support provided to these patients, early detection of their needs, connection with community care agents, monitoring of treatment adherence, and remote interventions targeted towards prevention of relapse.

ELIGIBILITY:
Inclusion Criteria:

Men & women,

1. age 18-60 ,
2. "Maccabi Health service" patients with diagnosis of: schizophrenia, Schizo - effective or Bipolar Dis.
3. Must have 30 days or more of hospitalization (during 3 years). Treated with psychiatric medication.
4. Living independently or with a help of a caregiver.
5. Is able to provide written informed consent.

Exclusion Criteria:

1. Violent, or suicidal.
2. Drug\ Alcohol, addiction,
3. End stage Disease (Cancer, ESRF act.)
4. Non - in depended and without Care giver/legal guardian

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
number of days of hospitalization | through study competion ,an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Asaf B Caspi, MD, Principal Investigator — Sheba Medical Center

IPD SHARING:
Plan to Share IPD: Yes